CLINICAL TRIAL: NCT00898352
Title: Phase III Radiation Therapy vs Pelvic Node Resection for Previously Untreated Invasive Squamous Cell Carcinoma of the Vulva With Positive Groin Nodes
Brief Title: Radiation Therapy or Surgery in Treating Patients With Previously Untreated Vulva Cancer With Positive Groin Lymph Nodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Philip J. DiSaia, Gynecologic Oncology Group
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000070950; GOG-37; GOG-7712
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2009-10

CONDITIONS: Vulvar Cancer
Keywords: stage III vulvar cancer; squamous cell carcinoma of the vulva
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: regional lymph node dissection
Radiation: radiation therapy

SUMMARY:
RATIONALE: Patient abstract not available

PURPOSE: Patient abstract not available

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of pelvic node resection vs. bilateral groin and pelvic node irradiation for invasive squamous cell carcinoma of the vulva in patients having positive groin nodes.

OUTLINE: Randomized study. Arm I: Surgery. Deep pelvic node dissection on sides containing positive nodes only. Arm II: Radiotherapy. Megavoltage (1 MeV or greater) to bilateral groin and pelvic nodes.

PROJECTED ACCRUAL: Anticipated annual accrual is approximately 200 patients, with an active phase estimated at 2.5-3 years. Protocol closed July 1984.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: See General Eligibility Criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 1990-11 (Actual)

PRIMARY OUTCOMES:
Recurrence rate
Survival rate
Subjective status on GOG performance scale
Time to recurrence
Survival time
Morbidity of treatment

CONTACTS AND LOCATIONS:
Overall Officials: George C. Lewis, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University

REFERENCES:
- [Result] Kunos C, Simpkins F, Gibbons H, Tian C, Homesley H. Radiation therapy compared with pelvic node resection for node-positive vulvar cancer: a randomized controlled trial. Obstet Gynecol. 2009 Sep;114(3):537-546. doi: 10.1097/AOG.0b013e3181b12f99. PMID 19701032
- [Result] Homesley HD, Bundy BN, Sedlis A, Adcock L. Radiation therapy versus pelvic node resection for carcinoma of the vulva with positive groin nodes. Obstet Gynecol. 1986 Dec;68(6):733-40. PMID 3785783